CLINICAL TRIAL: NCT06124105
Title: Can Urinary Partial Oxygen Pressure be an Indicator of Acute Kidney Injury in Patients With Sepsis?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Murat Bıçakcıoğlu, Principal Investigator, Inonu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MB2
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Acute Kidney Injury; Sepsis
Keywords: acute kidney injrury, sepsis, urine parcial oxygen pressure
MeSH Terms: conditions — Acute Kidney Injury; Sepsis | interventions — Blood Gas Analysis

STUDY DESIGN:
Intervention Model Description: study group: patients who develop aki in sepsis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- urine PO2 (Other)
  Interventions: Diagnostic Test: arterial blood gases

INTERVENTIONS:
Diagnostic Test: arterial blood gases — measurement of partial oxygen pressure in urine by arterial blood gas device

SUMMARY:
The ability of bladder urinary partial pressure, measured as a reflection of renal medullary oxygen tension, which is an indicator of the development of acute kidney injury (AKI), to predict the development of AKI at an early stage.

DETAILED DESCRIPTION:
Patients hospitalised in the intensive care unit with a diagnosis of sepsis will be followed up for the development of ABH. This follow-up will be performed for 5 days after hospitalisation. During this period, patients will be sampled for NGAL 5 times in total, once every day. PuO2 will be sampled daily to determine PuO2 and to observe the development of AKI, and in cases of hypotension where the mean arterial pressure falls below 65 mmHg or in cases of severe acidosis, extra will be sampled at least 5 times, once every day. PuO2 will be analysed in the blood gas device and PuO2 value will be recorded. For NGAL analysis, patient blood will be collected in ETDA tubes and stored at -80 °C until analysis. NGAL will then be measured by turbidimetric imminoassay method. The comorbidities of the patients will be questioned and recorded, the types and amounts of fluids taken, whether they received blood and blood products, and if so, which product and how much they received will be recorded. APACHI II score and SOFA scores of the patients at hospitalisation will be recorded. GCS, whether mechanical ventilation support is provided or not, if any, ventilation method, mode and ventilation parameters will be recorded. In addition to these, mean arterial pressure, pulse, temperature, SpO2, FiO2 values will be recorded clinically. Haemoglobin, haemotocrit, platelets, bun, creatinine, biluribins, liver function tests and arterial blood gas will be recorded in the laboratory. In addition, whether the patients have ARDS, whether they are receiving renal replacement therapy and if so, the prescription and ultrasonography findings will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to intensive care unit with sepsis

Exclusion Criteria:

* Causing an infection other than sepsis at the time of admission
* Acute renal failure at the time of admission
* Having a creatinine value above 1.5 mg/dL at the time of admission
* Previously known chronic renal failure or being on a routine dialysis programme (receiving renal replacement therapy)
* Having one kidney
* Having another known kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-03-06 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury | first 5 days
  urine partial oxygen pressure in arterial blood gases

SECONDARY OUTCOMES:
mortality | 28. days
  death rate

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Osawa EA, Cutuli SL, Bitker L, Canet E, Cioccari L, Iguchi N, Lankadeva YR, Eastwood GM, Evans RG, May CN, Bellomo R. Effect of Furosemide on Urinary Oxygenation in Patients with Septic Shock. Blood Purif. 2019;48(4):336-345. doi: 10.1159/000501512. Epub 2019 Jul 23. PMID 31336370
- [Background] Silverton NA, Lofgren LR, Hall IE, Stoddard GJ, Melendez NP, Van Tienderen M, Shumway S, Stringer BJ, Kang WS, Lybbert C, Kuck K. Noninvasive Urine Oxygen Monitoring and the Risk of Acute Kidney Injury in Cardiac Surgery. Anesthesiology. 2021 Sep 1;135(3):406-418. doi: 10.1097/ALN.0000000000003663. PMID 34329393
- [Background] Evans RG, Cochrane AD, Hood SG, Iguchi N, Marino B, Bellomo R, McCall PR, Okazaki N, Smith JA, Zhu MZ, Ngo JP, Noe KM, Martin A, Thrift AG, Lankadeva YR, May CN. Dynamic responses of renal oxygenation at the onset of cardiopulmonary bypass in sheep and man. Perfusion. 2022 Sep;37(6):624-632. doi: 10.1177/02676591211013640. Epub 2021 May 12. PMID 33977810